CLINICAL TRIAL: NCT00810381
Title: Ocular Hemodynamic Effects of Nitrovasodilators in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Hans-Georg Eichler, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-211097
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Glaucoma
Keywords: Nitrovasodilators; ONH blood flow; Choroidal blood flow; Nitroglycerin; Isosorbide Dinitrate; Sodium nitroprusside; Laser-Doppler Flowmetry; Regional Blood Flow
MeSH Terms: conditions — Glaucoma | interventions — Nitroglycerin; Isosorbide; Nitroprusside; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Nitroglycerin: (Perlinganit, Nycomet Heilmittelwerke, Vienna, Austria):
  0, 0.25, 0.5, 1, 1.5 and 2 µg/kg/min, each infusion step for 20 minutes
  Interventions: Drug: Nitroglycerin
- 2 (Active Comparator): Isosorbide-Dinitrate: (Isoket 0,1 %, Gebro Broschek, Fieberbrunn, Austria):
  0, 0.5, 1, 2, 4 and 6 µg/kg/min , each infusion step for 20 minutes
  Interventions: Drug: Isosorbide-Dinitrate
- 3 (Active Comparator): Sodium-Nitroprusside: (Nipruss, Sanol-Schwarz, Monheim, Germany):
  0, 0.25, 0.5, 1, 2 and 4 µg/kg/min, each infusion step for 20 minutes
  Interventions: Drug: Sodium-nitroprusside
- 4 (Placebo Comparator): Physiologic saline solution
  Interventions: Drug: Physiologic saline solution (control substance)

INTERVENTIONS:
Drug: Nitroglycerin — intravenous infusion; 0, 0.125, 0.25, 0.5, 1 and 2 µg/kg/min; 20 minutes per infusion step
  Arms: 1
Drug: Isosorbide-Dinitrate — intravenous infusion; 0, 0.5, 1, 2, 4, and 6 µg/kg/min; 20 minutes per infusion step
  Arms: 2
Drug: Sodium-nitroprusside — intravenous infusion; 0, 0.25, 0.5, 1, 2, and 4 µg/kg/min; 20 minutes per infusion step
  Arms: 3
Drug: Physiologic saline solution (control substance) — intravenous infusion, infusion period 120 minutes
  Arms: 4

SUMMARY:
Glaucoma, one of the most common causes of blindness, is associated with increased intraocular pressure (IOP) and optic nerve head ischemia. Nitrovasodilators are discussed in the treatment of glaucoma. Nitrates relax smooth muscle cells in the vasculature by liberating the vasodilator nitric oxide.

The IOP lowering potential and the vasodilator action in retinal and choroidal vessels of nitrates is still a matter of controversy. Previous studies on the ocular hemodynamic effects of nitrates showed partially contradicting results. In addition the IOP lowering effect of nitrates is still unclear. However, recent studies show that long acting nitrates may preserve optic nerve deterioration and visual field loss.

Therefore, the role of nitrovasodilators in control of ocular blood flow and intraocular pressure has to be elucidated. For this purpose the investigators plan to test the hypothesis that nitrovasodilators improve ocular blood supply to the optic nerve head at doses which do not affect systemic hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* History of migraine
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 1999-01; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
Optic disc blood flow (laser Doppler flowmetry) | in total 24x on 4 study days

SECONDARY OUTCOMES:
Intraocular pressure | in total 8x in 4 study days
Choroidal blood flow (laser Doppler flowmetry) | in total 24x on 4 study days
Fundus pulsation amplitude in the macula (laser interferometry) | in total 24x on 4 study days
Fundus pulsation amplitude in the optic disc (laser interferometry) | in total 24x on 4 study days
Blood pressure, pulse rate | on 4 study days

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Georg Eichler, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria